CLINICAL TRIAL: NCT07154589
Title: Effects of AbClo Fascial Approximation Device in Patients With Open Abdomen on Respiratory Mechanics (AbClo-Resp)
Brief Title: Effects of AbClo Fascial Approximation Device in Patients With Open Abdomen on Respiratory Mechanics
Acronym: AbClo-Resp
Status: Recruiting | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Laurent Brochard, Dr., Unity Health Toronto
Other Study IDs: 25-034
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Open Abdomen; Mechanical Ventilation
Keywords: open abdomen; mechanical ventilation; transpulmonary pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Abdominal fascial approximation device: All patients are already on the device before starting the study

SUMMARY:
Patients who underwent an abdominal surgery and had the abdomen remain open are called to have an "open abdomen". To limit the risk of further widening of their wounds, surgeons can use AbClo, which is a non-invasive abdominal binding device, to keep the abdominal wall together (i.e., approximate the fascia). However, as the device also compresses on the abdomen and adjacent lungs, this study aims:

* To assess whether the abdominal binding device causes changes in the pressure compressing the lungs, the lung volume, and the function of the lungs.
* To assess whether adjusting the breathing machine can mitigate such negative changes.

Participants will already be on the abdominal binding device when joining the study. Measurements on various aspects of the lung function (including its physical properties and capability to oxygenate the blood) will be done before and after adjustment of the abdominal binding device to the pressure (measured in the device itself) recommended by the manufacturer, as well as after the surgery to close the abdomen.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older
* Patients admitted to an ICU
* Patients with postoperative abdominal surgery with open abdomen
* Patients treated with AbClo device
* Patients intubated and mechanically ventilated
* Patients treated with intravenous sedation with a sedation-agitation scale score of 1-3

Exclusion Criteria:

* Transient criteria: Patients with severe hemodynamic instability, defined systolic blood pressure less than 75 mmHg or mean arterial pressure less than 60 mmHg despite vasopressor use
* Transient criteria: Patients with severe bleeding diathesis, defined as the latest platelet count less than 20 · 109/L, or the latest INR higher than 2.0
* Patients with concurrent injuries to upper gastrointestinal tract that would preclude esophageal balloon insertion
* Patients with bronchopleural fistula
* Patients with measured and uncontrolled increased intracranial pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted the ICU with open abdomen treated with AbClo device, and undergoing mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Changes in End-expiratory Transpulmonary Pressure | On the day of enrolment and on the day of surgery to close the abdomen
  Calculated by the difference between airway pressure and the value measured by an esophageal catheter at the end of expiration. Measurements are made once before the adjustment of the fascial approximation device to the optimal pressure, after the adjustment, and again after the surgery to close the abdomen.

SECONDARY OUTCOMES:
Changes in Lung Volume | On the day of enrolment
  Measured by a ventilator capable of measuring end-expiratory lung volume, using a breath-in-breath-out method. Measurements are made once before the adjustment of the fascial approximation device to the optimal pressure, and again after the adjustment.
Changes in oxygenation function | On the day of enrolment and on the day of surgery to close the abdomen
  Determined by the partial pressure of oxygen and PaO₂/FiO₂ ratio from arterial blood gas. Measurements are made once before the adjustment of the fascial approximation device to the optimal pressure, after the adjustment, and again after the surgery to close the abdomen.
Response in End-expiratory Transpulmonary Pressure to PEEP Increase | On the day of enrolment
  In participants with negative end-expiratory transpulmonary pressure with clinically set PEEP, under the supervision of the clinical team in the ICU, PEEP will be titrated up until until zero or positive values are restored. Responses to the titration will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The datasets generated and/or analyzed during the current study will not be publicly available due participant confidentiality, according to the REB, but will be available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Wauters J, Wilmer A, Valenza F. Abdomino-thoracic transmission during ACS: facts and figures. Acta Clin Belg. 2007;62 Suppl 1:200-5. PMID 17469720
- [Background] Regli A, Pelosi P, Malbrain MLNG. Ventilation in patients with intra-abdominal hypertension: what every critical care physician needs to know. Ann Intensive Care. 2019 Apr 25;9(1):52. doi: 10.1186/s13613-019-0522-y. PMID 31025221
- [Background] Beitler JR, Sarge T, Banner-Goodspeed VM, Gong MN, Cook D, Novack V, Loring SH, Talmor D; EPVent-2 Study Group. Effect of Titrating Positive End-Expiratory Pressure (PEEP) With an Esophageal Pressure-Guided Strategy vs an Empirical High PEEP-Fio2 Strategy on Death and Days Free From Mechanical Ventilation Among Patients With Acute Respiratory Distress Syndrome: A Randomized Clinical Trial. JAMA. 2019 Mar 5;321(9):846-857. doi: 10.1001/jama.2019.0555. PMID 30776290
- [Background] Yoshida T, Amato MBP, Grieco DL, Chen L, Lima CAS, Roldan R, Morais CCA, Gomes S, Costa ELV, Cardoso PFG, Charbonney E, Richard JM, Brochard L, Kavanagh BP. Esophageal Manometry and Regional Transpulmonary Pressure in Lung Injury. Am J Respir Crit Care Med. 2018 Apr 15;197(8):1018-1026. doi: 10.1164/rccm.201709-1806OC. PMID 29323931
- [Background] Naveed A, Martin ND, Bawazeer M, Jastaniah A, Rezende-Neto JB. Early placement of a non-invasive, pressure-regulated, fascial reapproximation device improves reduction of the fascial gap in open abdomens: a retrospective cohort study. Trauma Surg Acute Care Open. 2024 Oct 12;9(1):e001529. doi: 10.1136/tsaco-2024-001529. eCollection 2024. PMID 39411009
- [Background] Rezende-Neto JB, Camilotti BG. New non-invasive device to promote primary closure of the fascia and prevent loss of domain in the open abdomen: a pilot study. Trauma Surg Acute Care Open. 2020 Nov 11;5(1):e000523. doi: 10.1136/tsaco-2020-000523. eCollection 2020. PMID 33225070
- [Background] Diaz JJ Jr, Cullinane DC, Dutton WD, Jerome R, Bagdonas R, Bilaniuk JW, Collier BR, Como JJ, Cumming J, Griffen M, Gunter OL, Kirby J, Lottenburg L, Mowery N, Riordan WP Jr, Martin N, Platz J, Stassen N, Winston ES. The management of the open abdomen in trauma and emergency general surgery: part 1-damage control. J Trauma. 2010 Jun;68(6):1425-38. doi: 10.1097/TA.0b013e3181da0da5. PMID 20539186
- [Background] Roberts DJ, Leppaniemi A, Tolonen M, Mentula P, Bjorck M, Kirkpatrick AW, Sugrue M, Pereira BM, Petersson U, Coccolini F, Latifi R. The open abdomen in trauma, acute care, and vascular and endovascular surgery: comprehensive, expert, narrative review. BJS Open. 2023 Sep 5;7(5):zrad084. doi: 10.1093/bjsopen/zrad084. PMID 37882630
- [Background] Kreis BE, de Mol van Otterloo AJ, Kreis RW. Open abdomen management: a review of its history and a proposed management algorithm. Med Sci Monit. 2013 Jul 3;19:524-33. doi: 10.12659/MSM.883966. PMID 23823991
- [Background] Kirkpatrick AW, Roberts DJ, De Waele J, Jaeschke R, Malbrain ML, De Keulenaer B, Duchesne J, Bjorck M, Leppaniemi A, Ejike JC, Sugrue M, Cheatham M, Ivatury R, Ball CG, Reintam Blaser A, Regli A, Balogh ZJ, D'Amours S, Debergh D, Kaplan M, Kimball E, Olvera C; Pediatric Guidelines Sub-Committee for the World Society of the Abdominal Compartment Syndrome. Intra-abdominal hypertension and the abdominal compartment syndrome: updated consensus definitions and clinical practice guidelines from the World Society of the Abdominal Compartment Syndrome. Intensive Care Med. 2013 Jul;39(7):1190-206. doi: 10.1007/s00134-013-2906-z. Epub 2013 May 15. PMID 23673399
- [Background] Mahoney EJ, Bugaev N, Appelbaum R, Goldenberg-Sandau A, Baltazar GA, Posluszny J, Dultz L, Kartiko S, Kasotakis G, Como J, Klein E. Management of the open abdomen: A systematic review with meta-analysis and practice management guideline from the Eastern Association for the Surgery of Trauma. J Trauma Acute Care Surg. 2022 Sep 1;93(3):e110-e118. doi: 10.1097/TA.0000000000003683. Epub 2022 May 12. PMID 35546420